CLINICAL TRIAL: NCT05851729
Title: Effects of Kegal Exercises With and Without Postural Correction on Postpartum Pelvic Organ Prolapse in Primiparous Women
Brief Title: Kegal Exercises With and Without Postural Correction on Postpartum Pelvic Organ Prolapse in Primiparous Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0517
Record Dates: First submitted 2023-03-31; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kegal exercises with postural correction (Experimental)
  Interventions: Other: Kegal exercises with postural correction
- Kegal exercises without postural correction (Experimental)
  Interventions: Other: Kegal exercises without postural correction

INTERVENTIONS:
Other: Kegal exercises with postural correction — Kegal exercises with postural correction
  Arms: Kegal exercises with postural correction
Other: Kegal exercises without postural correction — Kegal exercises without postural correction
  Arms: Kegal exercises without postural correction

SUMMARY:
To study the effects of kegal exercises with and without postural correction on pelvic organ prolapse in primiparous women. Although pregnancy is a physiological process, it is associated with risk factors. These risk factors can put women at risk. One of the most common problems is pelvic floor muscle weakness, and this weakness of pelvic floor muscles causes many other problems, such as pelvic organ prolapse. Normal delivery (vaginal delivery) can cause laxity and weakness of ligaments such as the external urethral and pubourethral. Pelvic organs prolapse severely affects the quality of life of patients. Pelvic organ prolapse appears in women after vaginal delivery. Pelvic muscle training is a conservative treatment for many problems, including pelvic organ prolapse. However, the effects of pelvic floor muscle training for pelvic organ prolapse in primiparous women are controversial. This study is aimed at a systematic review of the effects of pelvic floor muscle training on pelvic organ prolapse in primiparous women.

DETAILED DESCRIPTION:
The design of this study will randomize controlled trial. Data will collect from the Settings of Jinnah Hospital Lahore, THQ Hospital Depalpur, and Al-Shifa Hospital Depalpur. The sample size for this study is 30 primiparous women. Participants will be screened for eligibility. Women will be randomly assigned to the training group, which conducts 12 weekly individual sessions. Outcomes will be assessed after the last session. The control group will receive kegal exercise after the initial assessment. Main outcome measures for this study include the symptoms pelvic floor impact questionnaire, the pelvic floor distress inventory questionnaire, and the pelvic organ prolapse quantification examination. The pelvic floor impact questionnaire will assess the lifelong impact of pelvic floor disorders on women.

A pelvic floor distress inventory questionnaire will assess distress caused by PFD (pelvic floor dysfunction).

ELIGIBILITY:
Inclusion Criteria:

* Primiparous,Age: 20-40,
* 6th to 8th week after delivery,
* Singleton baby vaginally fully term,
* Non instrumented birth of child,
* Grade 1 prolapse (5)

Exclusion Criteria:

* Women with Chronic Cough,
* Constipation,
* Previous Pelvic surgery,
* Pelvic malignancy,
* Genitourinary Infection

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-03 (Estimated); Study Completion 2023-06-03 (Estimated)

PRIMARY OUTCOMES:
Pelvic Floor Impact Questionnaire. (PFIQ-7) | 1st day
  The PFIQ is a patient report designed to assess life impact of pelvic floor disorders on women

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Mehjabeen, MS(WHPT), Principal Investigator — Riphah International University
Locations (1):
- Services Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sigurdardottir T, Steingrimsdottir T, Geirsson RT, Halldorsson TI, Aspelund T, Bo K. Postpartum pelvic organ prolapse and pelvic floor muscle training: secondary analysis of a randomized controlled trial of primiparous women. Int Urogynecol J. 2023 Jun;34(6):1319-1326. doi: 10.1007/s00192-023-05502-8. Epub 2023 Mar 30. PMID 36995416
- [Background] Artymuk NV, Khapacheva SY. Device-assisted pelvic floor muscle postpartum exercise programme for the management of pelvic floor dysfunction after delivery. J Matern Fetal Neonatal Med. 2022 Feb;35(3):481-485. doi: 10.1080/14767058.2020.1723541. Epub 2020 Feb 4. PMID 32019378